CLINICAL TRIAL: NCT01700127
Title: Predictors of Poor Immune Response to Rotavirus Vaccine in Infants
Acronym: PPIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: Christian Medical College, Vellore, India (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SAS/RCN/201208
Record Dates: First submitted 2012-09-28; First posted 2012-10-04 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Innate Immune Response
Keywords: immune response; infants; rotavirus vaccine
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breastfeeding (Other): Breastfeeding Encouraged
  Interventions: Other: Breastfeeding
- Breastfeeding Withheld (Active Comparator): Breastfeeding Withheld
  Interventions: Other: Breastfeeding

INTERVENTIONS:
Other: Breastfeeding — breastfeeding encouraged versus withheld

SUMMARY:
This will be a randomized study with the primary objective of assessing the impact of withholding versus encouraging breastfeeding on the immunogenicity of Rotarix® in infants.

Enrolled subjects will all be administered Rotarix®, at ages 6 to 7 weeks, and at10 -14 weeks. The subjects will be randomized into one of the two study arms. In one of the group caregivers will be advised to breastfeed immediately prior to and after each dose of the vaccine while in the other group caregivers will be advised to withhold breastfeeding for 30 minutes before and after each dose of the vaccine. The other childhood vaccines i.e. OPV and Pentavalent will be administered at least 30 minutes after administration of Rotarix®, The enrolled subjects will be followed up for 4 weeks after the 2nd dose of Rotarix®.

DETAILED DESCRIPTION:
Infants ≤7 weeks and pregnant women will be identified through a household survey.Families of infants aged 6-7 weeks will be called to the study clinic for consenting, screening and enrollment.All enrolled subjects will be administered 2 doses of Rotarix® at 6 to 7 weeks and at 10-14 weeks of age. Other childhood vaccines will also be offered.

At enrollment, a blood specimen and breast milk specimen will be obtained from the mother and a blood, salivary and stool specimens will be obtained from the subject before administering the Rotarix® vaccine.

At the time of the 2nd administration, a breast milk specimen will be obtained from the mother and a salivary specimen will be obtained from the subject before administering the Rotarix® vaccine. At 28 days (±) 5 after the 2nd dose of Rotarix® vaccine, a blood, salivary and stool specimen will be obtained from the subject.

Whenever the family comes to the study clinic at 6-7 weeks, consent will be administered and a clinical examination conducted.If the family is willing for the mother and the child to be part of the study and the child meets the eligibility criteria, the child will be enrolled.

Depending on the group allocation the mothers will be advised to withhold or encourage breastfeeding for 30 minutes before and after receipt of Rotarix®.

subjects will be observed for 30 minutes after receipt of the vaccines to assess for immediate adverse events.

All minor illnesses that do not require hospital referral will be managed by the study physician using current practices.

All hospitalizations and deaths will be reported and reviewed by an Independent Safety Monitor.

ELIGIBILITY:
Inclusion Criteria:

1. At least one parent(s) or legally acceptable representative's consent for participation and are able to understand study procedures
2. Subjects aged 6 to 7 weeks at recruitment
3. No plans to move in the next 4 months
4. Weight for age not ≤ -3 SD of WHO child growth standards

Exclusion Criteria:

1. Infant not breastfed
2. Administration of rotavirus vaccine in the past
3. Known immunodeficiency disease, including HIV infection in the subject or the mother
4. Known chronic enteric disease
5. Diarrhea on the day of enrollment (temporary exclusion)
6. Any illness requiring hospitalization (temporary exclusion)
7. Any other conditions which in the judgment of the investigator warrant exclusion (e.g. no exclusion criteria but seems 'ill', investigators suspects neglect)

Ages: 6 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who seroconvert as measured by a 4-fold rise in serum anti-VP6 IgA antibodies between baseline and 4 weeks after the second dose of Rotarix®. | 14-18 weeks of age

SECONDARY OUTCOMES:
Concentration of anti-VP6 antibodies in saliva of subjects before the first and second dose of Rotarix®. Proportion of subjects with enteric pathogens detected in stools. Vitamin D status of subjects enrolled in the study. | 14-18 weeks of age

OTHER OUTCOMES:
Concentration of anti-VP6 antibodies in subjects and maternal serum at baseline and in subjects 4 weeks after the second dose of Rotarix®. Geometric mean titers of anti-VP6 IgG antibodies in maternal serum at baseline | upto 14-18 weeks of age

CONTACTS AND LOCATIONS:
Overall Officials: Temsunaro R Chandola, MBBS MSc Epi, Principal Investigator — Research Scientist, SAS; Nita Bhandari, MBBS, PhD, Principal Investigator — Joint Director, SAS; Sunita Taneja, MBBS, PhD, Principal Investigator — Research Coordinator, SAS; Gagandeep Kang, MD PhD FRCPath, Principal Investigator — Professor and Head,The Wellcome Trust Research Laboratory,Christian Medical College; Tor A Strand, MD, PhD, Principal Investigator — Adjunct Professor, CIH
Locations (1):
- Centre for Health Research and Development Society for Applied Studies, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Rongsen-Chandola T, Strand TA, Goyal N, Flem E, Rathore SS, Arya A, Winje BA, Lazarus R, Shanmugasundaram E, Babji S, Sommerfelt H, Vainio K, Kang G, Bhandari N. Effect of withholding breastfeeding on the immune response to a live oral rotavirus vaccine in North Indian infants. Vaccine. 2014 Aug 11;32 Suppl 1:A134-9. doi: 10.1016/j.vaccine.2014.04.078. PMID 25091668
- [Derived] Rongsen-Chandola T, Winje BA, Goyal N, Rathore SS, Mahesh M, Ranjan R, Arya A, Rafiqi FA, Bhandari N, Strand TA. Compliance of mothers following recommendations to breastfeed or withhold breast milk during rotavirus vaccination in North India: a randomized clinical trial. Trials. 2014 Jun 28;15:256. doi: 10.1186/1745-6215-15-256. PMID 24976452